CLINICAL TRIAL: NCT04908930
Title: Community-Engaged Sport Safety - Aim 1 and Aim 3
Brief Title: Evidence-based Intervention for Improved Head Impact Safety in Youth Football - Aim 1 and Aim 3
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Supportive Care
Other Study IDs: IRB00067187; K25HD101686 (NIH)
Record Dates: First submitted 2021-05-17; First posted 2021-06-01 (Actual); Results first posted 2025-02-27 (Actual); Last update posted 2025-02-27 (Actual); Status verified 2023-03

CONDITIONS: Head Injury; Sport Injury
Keywords: Sport Safety; Youth Football; Head Impact Exposure
MeSH Terms: conditions — Craniocerebral Trauma

STUDY DESIGN:
Intervention Model Description: All interested football players on the 2 teams will be enrolled; will be randomly selected for instrumentation with head impact sensors using a random numbers table. Athletes on these teams will follow their coach prescribed practice structure.
  Two additional youth football teams at the middle school level will be recruited to pilot test the intervention developed in this study. All interested athletes on these teams will be enrolled; will be randomly selected for instrumentation with head impact sensors using a random numbers table.
  Enrolled athletes will wear head impact sensors embedded in a custom mouthpiece that will be used to collect head impact exposure in conjunction with on-field video data for the season.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (5):
- Unexposed practice group- Aim 1 (No Intervention): Data from an unexposed sample (football players practicing as they would otherwise).
- On-field activity group - Aim 3 (Experimental): Athletes of two new teams at the middle school level to pilot the practice structure intervention and continuously monitor on-field activity with head impact sensors to evaluate the feasibility, acceptability, and sustainability of the practice structure
  Interventions: Behavioral: On-field activity group - Aim 3
- Unexposed practice group- Aim 1 Stakeholders (No Intervention): Stakeholders (parents, coaches, league officials) participated in guided discussions using an audit and feedback approach (sharing biomechanical data with the stakeholders) and semi-structured focus groups with the coaches and parents of the participating teams. Also, key informant interviews with league officials were used to assess the awareness and receptivity to creating a safer practice structure.
- On-field activity group - Aim 3 Stakeholders (Experimental): coaches pilot tested the COACH program
  Interventions: Behavioral: On-field activity group - Aim 3
- Unexposed Practice Group - Other Aim Stakeholders (No Intervention): Parent and organizational leader stakeholders (unexposed to intervention) participated in guided discussions about safety and biomechanics in youth football

INTERVENTIONS:
Behavioral: On-field activity group - Aim 3 — Athletes of two new teams at the middle school level to pilot the practice structure intervention and continuously monitor on-field activity with head impact sensors to evaluate the feasibility, acceptability, and sustainability of the practice structure
  Arms: On-field activity group - Aim 3; On-field activity group - Aim 3 Stakeholders

SUMMARY:
Two middle school (ages 11-14) football teams will be in Aim 1 of this study. All interested athletes on these teams will be invited to voluntarily participate in biomechanical data collection; of those enrolled, 15-20 per team will be randomly selected for instrumentation with head impact sensors. In aim 3, two youth football teams at the middle school level will be recruited to pilot an intervention developed this study. The football coaches of each team will be prospectively recruited and enrolled. All interested athletes on these teams will be enrolled; of those enrolled, 15-20 per team will be randomly selected for instrumentation with head impact sensors. Baseline and post-season neurocognitive data will be collected.

DETAILED DESCRIPTION:
This study hypothesizes that (a) determinants at the individual (athlete), interpersonal (team & coach), and community levels (built & social environment) of the social ecological model may be identified and targeted to reduce head impact exposure in youth football practices, and (b) an evidence-based strategy to reduce head impact exposure in practices may be developed and pilot tested using a community-engaged approach.

ELIGIBILITY:
Inclusion Criteria:

* All athletes participating on the prospective teams will be eligible for the study, including those with braces longer than 6 months.

Exclusion Criteria:

* Athletes will be excluded from participation if they have had braces less than 6 months, or have dental appliances that may impede the fit of the mouthpiece device (e.g., Herbst Appliance).

Ages: 11 Years to 14 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 106 (Actual)
Dates: Start 2021-07-08 (Actual); Primary Completion 2023-10-22 (Actual); Study Completion 2023-11-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jill Urban, PhD, MPH, Principal Investigator — Wake Forest Health Sciences
Locations (1):
- Wake Forest Health Sciences, Winston-Salem, North Carolina, United States

IPD SHARING:
Plan to Share IPD: Yes
Participant Data and Study Protocol
Supporting Information: Study Protocol
Time Frame: Beginning 9 months and ending 36 months following article publication
Access Criteria: Individual participant data (IPD) collected in this study be shared using the Federal Interagency Traumatic Brain Injury Research (FITBIR) informatics system. The National Institute of Health FITBIR database is a data sharing resource for the Traumatic Brain Injury imaging research field. Data sharing forms will be used to upload biomechanical data and associated metadata according to the The National Institute of Neurological Disorders and Stroke Department of Defense (NINDS/DoD) Biomechanical Devices in TBI Common Data Elements (CDE). All data summarized in publications will also be made available upon email request to the study Principal Investigator and upon completion of a data-sharing agreement.

REFERENCES:
- [Derived] Urban JE, Moore JB, Marks ME, Holcomb TD, Patterson R, McCoy A, Miles CM, Stitzel JD, Foley KL. Protocol for COACH, an evidence-based intervention for improved head impact safety in youth American football developed using a community-engaged approach. Contemp Clin Trials Commun. 2024 Sep 17;42:101371. doi: 10.1016/j.conctc.2024.101371. eCollection 2024 Dec. PMID 39351080

RESULTS

PARTICIPANT FLOW:
Groups:
- Unexposed Practice Group- Aim 1 (Stakeholders): Coach stakeholders (unexposed to intervention) participated in guided discussions about safety and biomechanics in youth football
- On-field Activity Group - Aim 3 (Stakeholders): Coach stakeholders pilot tested the intervention
- Unexposed Practice Group - Other Stakeholders: Parent and organizational leader stakeholders (unexposed to intervention) participated in discussions about safety and biomechanics in youth football. Did not participate in the biomechanical and neurocognitive assessments in other arms. No outcomes associated with this arm.
Period: Overall Study
Arm/Group | Unexposed Practice Group- Aim 1 | On-field Activity Group - Aim 3 | Unexposed Practice Group- Aim 1 (Stakeholders) | On-field Activity Group - Aim 3 (Stakeholders) | Unexposed Practice Group - Other Stakeholders
Started | 36 | 34 | 6 | 12 | 18
Completed | 30 | 25 | 6 | 12 | 18
Not Completed | 6 | 9 | 0 | 0 | 0
Not completed — Lost to Follow-up | 1 | 1 | 0 | 0 | 0
Not completed — hardware in mouth | 1 | 1 | 0 | 0 | 0
Not completed — wrong team | 1 | 0 | 0 | 0 | 0
Not completed — quit team | 2 | 4 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 1 | 2 | 0 | 0 | 0
Not completed — parent not liking program | 0 | 1 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Unexposed Practice Group- Aim 1 Stakeholders: Coach stakeholders (unexposed to intervention) participated in guided discussions about safety and biomechanics in youth football
- On-field Activity Group - Aim 3 Stakeholders: Coach stakeholders pilot tested the intervention
- Total: Total of all reporting groups
Arm/Group | Unexposed Practice Group- Aim 1 | On-field Activity Group - Aim 3 | Unexposed Practice Group- Aim 1 Stakeholders | On-field Activity Group - Aim 3 Stakeholders | Unexposed Practice Group - Other Aim Stakeholders | Total
Number analyzed (Participants) | 36 | 34 | 6 | 12 | 18 | 106
Age, Continuous [Mean (Standard Deviation); unit: years] | 12.4 (0.55) | 12.5 (0.82) | 33.5 (5.2) | 34.5 (6.7) | 39.0 (6.7) | 12.4 (0.70)
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0 | 9 | 9
  Male | 36 | 34 | 6 | 12 | 8 | 96
  Unknown | 0 | 0 | 0 | 0 | 1 | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4 | 7 | 0 | 0 | 1 | 12
  Not Hispanic or Latino | 31 | 23 | 5 | 12 | 16 | 87
  Unknown or Not Reported | 1 | 4 | 1 | 0 | 1 | 7
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 25 | 11 | 4 | 9 | 10 | 59
  White | 6 | 15 | 1 | 1 | 6 | 29
  More than one race | 3 | 4 | 0 | 1 | 1 | 9
  Unknown or Not Reported | 2 | 4 | 1 | 1 | 1 | 9

OUTCOME MEASURES:

1. Primary Outcome: Number of Head Impacts
Description: Head impact data will be transformed to the head center of gravity using Matlab (Mathworks, Inc., Natick, MA) and quantified for practice sessions.
Time Frame: Month 3
Population: Missing participants-- Unexposed practice group: 1 incompatible with mouthpiece, 1 quit team before contact, and 1 did not attend practice sessions.
  On-Field activity group: 1 incompatible with mouthpiece, 2 quit team before contact, 2 didn't like mouthpiece fit
Measure: Mean (Standard Deviation); unit: total number of practice impacts
Arm/Group | Unexposed Practice Group- Aim 1 | On-field Activity Group - Aim 3
Number analyzed (Participants) | 33 | 29
total number of practice impacts | 100.24 (81.06) | 50.27 (39.57)

2. Primary Outcome: Number of Impacts Per Player Per Minute
Description: Head impact data will be transformed to the head center of gravity using Matlab (Mathworks, Inc., Natick, MA) and quantified for practice sessions. Number of impacts per player per minute
Time Frame: Month 3
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: impacts per player per minute
Arm/Group | Unexposed Practice Group- Aim 1 | On-field Activity Group - Aim 3
Number analyzed (Participants) | 33 | 29
impacts per player per minute | 0.047 (0.03) | 0.026 (0.02)

3. Primary Outcome: Mean Number of Impacts Per Athlete Per Practice
Description: as for outcome 1
Time Frame: Month 3
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Impacts per athlete per practice
Arm/Group | Unexposed Practice Group- Aim 1 | On-field Activity Group - Aim 3
Number analyzed (Participants) | 33 | 29
Impacts per athlete per practice | 4.75 (3.35) | 2.74 (2.03)

4. Primary Outcome: 95th Percentile Number of Impacts Per Athlete Per Practice
Description: as for outcome 1
Time Frame: Month 3
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Impacts/Athlete/ Practice
Arm/Group | Unexposed Practice Group- Aim 1 | On-field Activity Group - Aim 3
Number analyzed (Participants) | 33 | 29
Impacts/Athlete/ Practice | 15.12 (10.73) | 10.12 (5.95)

5. Primary Outcome: Median Linear Acceleration (g)
Description: Head impact data will be transformed to the head center of gravity using Matlab (Mathworks, Inc., Natick, MA) in terms of median linear acceleration.
Time Frame: Month 3
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: g
Arm/Group | Unexposed Practice Group- Aim 1 | On-field Activity Group - Aim 3
Number analyzed (Participants) | 33 | 29
g | 9.63 (2.05) | 12.7 (3.74)

6. Primary Outcome: Median Rotational Acceleration
Description: Head impact data will be transformed to the head center of gravity using Matlab (Mathworks, Inc., Natick, MA) in terms of median rotational acceleration.
Time Frame: Month 3
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: rad/s^2
Arm/Group | Unexposed Practice Group- Aim 1 | On-field Activity Group - Aim 3
Number analyzed (Participants) | 33 | 29
rad/s^2 | 722.03 (295.31) | 1035.21 (451.41)

7. Primary Outcome: Median Rotational Velocity
Description: Head impact data will be transformed to the head center of gravity using Matlab (Mathworks, Inc., Natick, MA) in terms of median rotational velocity.
Time Frame: Month 3
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: rad/s
Arm/Group | Unexposed Practice Group- Aim 1 | On-field Activity Group - Aim 3
Number analyzed (Participants) | 33 | 29
rad/s | 9.03 (2.25) | 10.28 (3.25)

8. Primary Outcome: 95th Percentile Linear Acceleration (g)
Description: Head impact data will be transformed to the head center of gravity using Matlab (Mathworks, Inc., Natick, MA) in terms of 95th percentile linear acceleration.
Time Frame: Month 3
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: g
Arm/Group | Unexposed Practice Group- Aim 1 | On-field Activity Group - Aim 3
Number analyzed (Participants) | 33 | 29
g | 25.8 (6.83) | 31.86 (10.46)

9. Primary Outcome: 95th Percentile Rotational Acceleration
Description: Head impact data will be transformed to the head center of gravity using Matlab (Mathworks, Inc., Natick, MA) in terms of 95th percentile rotational acceleration.
Time Frame: Month 3
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: rad/s^2
Arm/Group | Unexposed Practice Group- Aim 1 | On-field Activity Group - Aim 3
Number analyzed (Participants) | 33 | 29
rad/s^2 | 2013.18 (1014.19) | 2928.97 (1340.6)

10. Primary Outcome: 95th Percentile Rotational Velocity
Description: Head impact data will be transformed to the head center of gravity using Matlab (Mathworks, Inc., Natick, MA) in terms of 95th percentile rotational velocity.
Time Frame: Month 3
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: rad/s
Arm/Group | Unexposed Practice Group- Aim 1 | On-field Activity Group - Aim 3
Number analyzed (Participants) | 33 | 29
rad/s | 17.19 (2.89) | 21.21 (5.24)

11. Secondary Outcome: Feasibility of Intervention Measure (FIM)
Description: Perceived feasibility - higher values denote better feasibility - total range 0 - 5; 1, completely disagree; 5, completely agree - higher scores denote more possibility and agreeability to Intervention
Time Frame: Month 3
Population: No data collected for this outcome for the Unexposed Practice Group Stakeholders.
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Unexposed Practice Group-Stakeholders Aim 1: Coach stakeholders (unexposed to intervention) participated in guided discussions about safety and biomechanics in youth football
Arm/Group | Unexposed Practice Group-Stakeholders Aim 1 | On-field Activity Group - Aim 3 Stakeholders
Number analyzed (Participants) | 6 | 12
score on a scale | 4.75 (0.18) | 4.41 (0.54)

12. Secondary Outcome: Acceptability of Intervention Measure (AIM)
Description: total range 0 - 5 higher values denote better acceptability of the intervention (higher scores are better)
Time Frame: Month 3
Population: No data collected for this outcome for the Unexposed Practice Group Stakeholders.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Unexposed Practice Group- Aim 1 Stakeholders | On-field Activity Group - Aim 3 Stakeholders
Number analyzed (Participants) | 6 | 12
score on a scale | 5 (0) | 4.54 (0.5)

13. Secondary Outcome: Percentage of Practices the Intervention Was Implemented as Prescribed
Description: The intervention was prescribed to the North Carolina High School Athletic Association guidelines for contact in football practices, which limits teams to 15 minutes of live action contact per week. The percentage of practices the intervention was implemented as prescribed was monitored. An implementation score of 2 was given for adequate implementation (<15 minutes), 1 was given for partial implementation (<30 minutes), and 0 was given if live action contact exceeded 30 minutes for each practice. The percentage was calculated as the summed score for the season, divided by the maximum possible score across intervention teams.
Time Frame: Month 3
Population: Unexposed Practice Group- Aim 1 was not assessed for this measure because there is no intervention in that group.
  Therefore, unexposed practice group number analyzed value is zero. Missing participants--On-Field activity group: 1 incompatible with mouthpiece, 2 quit team before contact, 2 didn't like mouthpiece fit
Measure: Number; unit: percentage
Units Other Than Participants: Teams
Arm/Group | Unexposed Practice Group- Aim 1 | On-field Activity Group - Aim 3
Number analyzed (Participants) | 0 | 29
Number analyzed (Teams) | 0 | 2
percentage |  | 41.7

14. Secondary Outcome: Number Changes to the Intervention
Description: Adaptations to the intervention will be tracked as the number of changes to the intervention during the football season. Coach initiated adaptions will be tracked via visual observation. Adaptations advised by the stakeholder team will be tracked via meeting notes.
Time Frame: Month 3
Population: as for outcome 13
Measure: Number; unit: number of adaptations
Units Other Than Participants: teams
Arm/Group | Unexposed Practice Group- Aim 1 | On-field Activity Group - Aim 3
Number analyzed (Participants) | 0 | 29
Number analyzed (teams) | 0 | 2
number of adaptations |  | 0

15. Secondary Outcome: Verbal Memory (ImPACT) Immediate Post-Concussion Assessment and Cognitive Testing
Description: ImPACT is a computerized neuropsychological test battery. Participants will complete a pre-season baseline assessment which will be compared to post-season assessment scores - 0-100; higher scores are better
Time Frame: Baseline
Population: Missing participants-- Unexposed Group: 1 athlete did not complete data collection due to hardware in mouth (incompatible with mouthpiece) On-field Activity Group: 1 athlete did not have complete data collection due to hardware in mouth (incompatible with mouthpiece); 1 athlete did not attend baseline testing, and 3 athletes joined the study after the start of contact.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Unexposed Practice Group- Aim 1 | On-field Activity Group - Aim 3
Number analyzed (Participants) | 35 | 29
score on a scale | 74.57 (14.2) | 79.10 (11.18)

16. Secondary Outcome: Visual Memory Composite Score (ImPACT) Immediate Post-Concussion Assessment and Cognitive Testing
Description: as for outcome 15
Time Frame: Baseline
Population: as for outcome 15
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Unexposed Practice Group- Aim 1 | On-field Activity Group - Aim 3
Number analyzed (Participants) | 35 | 29
score on a scale | 63.77 (14.87) | 69.79 (13.24)

17. Secondary Outcome: (ImPACT) Immediate Post-Concussion Assessment and Cognitive Testing - Visual Motor Composite Score
Description: as for outcome 15
Time Frame: Baseline
Population: as for outcome 15
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Unexposed Practice Group- Aim 1 | On-field Activity Group - Aim 3
Number analyzed (Participants) | 35 | 29
score on a scale | 27.61 (7.82) | 27.87 (6.22)

18. Secondary Outcome: (ImPACT) Immediate Post-Concussion Assessment and Cognitive Testing - Reaction Time Composite Score
Description: ImPACT is a computerized neuropsychological test battery. Participants will complete a pre-season baseline assessment which will be compared to post-season assessment scores - 0-1; lower scores are better
Time Frame: Baseline
Population: as for outcome 15
Measure: Mean (Standard Deviation); unit: milliseconds
Arm/Group | Unexposed Practice Group- Aim 1 | On-field Activity Group - Aim 3
Number analyzed (Participants) | 35 | 29
milliseconds | 0.76 (0.11) | 0.72 (0.10)

19. Secondary Outcome: (ImPACT) Immediate Post-Concussion Assessment and Cognitive Testing - Impulse Control Composite Score
Description: ImPACT is a computerized neuropsychological test battery. Participants will complete a pre-season baseline assessment which will be compared to post-season assessment scores. Impulse control is a measure of errors on testing and is useful in determining test validity. This score indicates the sum of errors committed during different phases of the test - 0-40; lower scores are better
Time Frame: Baseline
Population: as for outcome 15
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Unexposed Practice Group- Aim 1 | On-field Activity Group - Aim 3
Number analyzed (Participants) | 35 | 29
score on a scale | 12.17 (11.44) | 11.17 (7.18)

20. Secondary Outcome: Flanker - National Institutes of Health (NIH) Toolbox Flanker Inhibitory Control and Attention Test Score
Description: Participants will complete a preseason baseline assessment which will be compared to post-season assessment scores - 70-120; higher scores are better
Time Frame: Baseline
Population: as for outcome 15
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Unexposed Practice Group- Aim 1 | On-field Activity Group - Aim 3
Number analyzed (Participants) | 35 | 29
score on a scale | 93.2 (20.98) | 91.24 (16.77)

21. Secondary Outcome: Flanker - National Institutes of Health (NIH) Toolbox Flanker Inhibitory Control and Attention Test Score
Description: as for outcome 20
Time Frame: Month 3
Population: Missing from each group-- Unexposed practice group: 1 was incompatible with mouthpiece, 1 had season-ending injury, 3 quit team, 1 did not like mouthpiece, and 5 did not return for testing.
  On-field activity group: 1 incompatible with mouthpiece, 1 athlete's parent withdrew consent, 4 quit the team, 2 did not like mouthpiece, 1 did not attend baseline testing, 3 joined study after start of contact during season, 1 didn't return for post-season testing.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Unexposed Practice Group- Aim 1 | On-field Activity Group - Aim 3
Number analyzed (Participants) | 25 | 21
score on a scale | 100.80 (18.67) | 98.19 (22.26)

22. Secondary Outcome: NIH Toolbox List Sorting Working Memory Test Score
Description: Participants will complete a preseason baseline assessment which will be compared to post-season assessment scores - List Sorting Working Memory; the score range is 50-150 - higher scores are better
Time Frame: Baseline
Population: as for outcome 15
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Unexposed Practice Group- Aim 1 | On-field Activity Group - Aim 3
Number analyzed (Participants) | 35 | 29
score on a scale | 105.77 (14.82) | 103.76 (15.99)

23. Secondary Outcome: NIH Toolbox List Sorting Working Memory Test Score
Description: as for outcome 22
Time Frame: Month 3
Population: as for outcome 21
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Unexposed Practice Group- Aim 1 | On-field Activity Group - Aim 3
Number analyzed (Participants) | 25 | 21
score on a scale | 128.28 (14.58) | 104.95 (17.45)

24. Secondary Outcome: NIH Toolbox Picture Vocabulary Test Score
Description: Participants will complete a preseason baseline assessment which will be compared to post-season assessment scores - Picture Vocabulary - 70-120; higher scores are better
Time Frame: Baseline
Population: as for outcome 15
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Unexposed Practice Group- Aim 1 | On-field Activity Group - Aim 3
Number analyzed (Participants) | 35 | 29
score on a scale | 91.89 (16.06) | 92.28 (11.68)

25. Secondary Outcome: NIH Toolbox Picture Sequence Memory Test Score
Description: Participants will complete a preseason baseline assessment which will be compared to post-season assessment scores - Picture Sequence Memory - 70-120; higher scores are better
Time Frame: Baseline and month 3
Population: Data not collected from any athletes for this outcome because this task was inadvertently not included in the testing protocol.
Arm/Group | Unexposed Practice Group- Aim 1 | On-field Activity Group - Aim 3
Number analyzed (Participants) | 0 | 0

26. Secondary Outcome: NIH Toolbox Picture Vocabulary Test Score
Description: as for outcome 24
Time Frame: Month 3
Population: as for outcome 21
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Unexposed Practice Group- Aim 1 | On-field Activity Group - Aim 3
Number analyzed (Participants) | 25 | 21
score on a scale | 92.52 (14.95) | 91.29 (11.18)

27. Secondary Outcome: Rey Auditory Verbal Learning Test Score (RAVLT)
Description: The RAVLT assesses verbal learning ability - A series of 15 words is presented to the participant 3 times via audio recording for standardization, and answers are recorded - Participants will complete a preseason baseline assessment which will be compared to post-season assessment scores - 0-45; higher scores are better
Time Frame: Baseline
Population: as for outcome 15
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Unexposed Practice Group- Aim 1 | On-field Activity Group - Aim 3
Number analyzed (Participants) | 35 | 29
score on a scale | 22.06 (6.29) | 23.28 (6.47)

28. Secondary Outcome: Rey Auditory Verbal Learning Test Score (RAVLT)
Description: as for outcome 27
Time Frame: Month 3
Population: as for outcome 21
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Unexposed Practice Group- Aim 1 | On-field Activity Group - Aim 3
Number analyzed (Participants) | 25 | 21
score on a scale | 29.76 (5.58) | 25.71 (7.44)

29. Secondary Outcome: Postural Control - Anterior-Posterior Postural Sway Score
Description: Participants will complete two 30-second trials (one with eyes opened, one with eyes closed) while standing on a force plate - Participants will complete a preseason baseline assessment which will be compared to post-season assessment scores - 0-50; lower scores are better
Time Frame: Baseline and month 3
Reporting Status: Not Posted

30. Secondary Outcome: Postural Control - Medial-Lateral Postural Sway Score
Description: as for outcome 29
Time Frame: Baseline and month 3
Reporting Status: Not Posted

31. Secondary Outcome: Postural Control - Maximum Path Velocity Score
Description: Participants will complete two 30-second trials (one with eyes opened, one with eyes closed) while standing on a force plate - Participants will complete a preseason baseline assessment which will be compared to post-season assessment scores - 0-10; lower scores are better
Time Frame: Baseline and month 3
Reporting Status: Not Posted

32. Secondary Outcome: Postural Control - Center of Pressure Area Score
Description: Participants will complete two 30-second trials (one with eyes opened, one with eyes closed) while standing on a force plate - Participants will complete a preseason baseline assessment which will be compared to post-season assessment scores - 0-20; lower scores are better
Time Frame: Baseline and month 3
Reporting Status: Not Posted

33. Secondary Outcome: Vestibular/Ocular Motor Screening (VOMS) - Smooth Pursuits
Description: The participant will be asked to focus on a small target that will be moved horizontally and vertically. The participant will report any symptoms (i.e., headache, dizziness, nausea, fogginess) after the task is complete. Symptoms reported range on a scale from 0-10; lower scores are better.
Time Frame: Baseline
Population: as for outcome 15
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Unexposed Practice Group- Aim 1 | On-field Activity Group - Aim 3
Number analyzed (Participants) | 35 | 29
score on a scale | 0.25 (0.76) | 0.11 (0.39)

34. Secondary Outcome: Vestibular/Ocular Motor Screening (VOMS) - Smooth Pursuits
Description: as for outcome 33
Time Frame: Month 3
Population: as for outcome 21
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Unexposed Practice Group- Aim 1 | On-field Activity Group - Aim 3
Number analyzed (Participants) | 25 | 21
score on a scale | 0.15 (0.49) | 0.06 (0.27)

35. Secondary Outcome: Vestibular/Ocular Motor Screening (VOMS) - Convergence
Description: The participant will be asked to focus on a small target and slowly bring it to the tip of their nose until two distinct images of the target are seen. The participant will complete this three times. The participant will report any symptoms (i.e., headache, dizziness, nausea, fogginess) after the task is complete. Symptoms reported range on a scale from 0-10; lower scores are better.
Time Frame: Month 3
Population: as for outcome 21
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Unexposed Practice Group- Aim 1 | On-field Activity Group - Aim 3
Number analyzed (Participants) | 25 | 21
score on a scale | 0.13 (0.39) | 0.10 (0.31)

36. Secondary Outcome: Vestibular/Ocular Motor Screening (VOMS) - Horizontal Saccades
Description: The participant will be asked to focus on two small targets that are horizontally aligned, moving their eyes quickly from one target to the other. The participant will report any symptoms (i.e., headache, dizziness, nausea, fogginess) after the task is complete. Symptoms reported range on a scale from 0-10; lower scores are better.
Time Frame: Baseline
Population: as for outcome 15
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Unexposed Practice Group- Aim 1 | On-field Activity Group - Aim 3
Number analyzed (Participants) | 35 | 29
score on a scale | 0.30 (0.78) | 0.12 (0.36)

37. Secondary Outcome: Vestibular/Ocular Motor Screening (VOMS) - Horizontal Saccades
Description: as for outcome 36
Time Frame: Month 3
Population: as for outcome 21
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Unexposed Practice Group- Aim 1 | On-field Activity Group - Aim 3
Number analyzed (Participants) | 25 | 21
score on a scale | 0.16 (0.48) | 0.10 (0.30)

38. Secondary Outcome: Vestibular/Ocular Motor Screening (VOMS) - Convergence
Description: as for outcome 35
Time Frame: Baseline
Population: as for outcome 15
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Unexposed Practice Group- Aim 1 | On-field Activity Group - Aim 3
Number analyzed (Participants) | 35 | 29
score on a scale | 0.35 (0.85) | 0.09 (0.31)

39. Secondary Outcome: Vestibular/Ocular Motor Screening (VOMS) - Visual Motion Sensitivity
Description: The participant will be asked to focus on a small target that they are holding still while rotating their torso from side to side. The participant will report any symptoms (i.e., headache, dizziness, nausea, fogginess) after the task is complete. Symptoms reported range on a scale from 0-10; lower scores are better.
Time Frame: Baseline
Population: as for outcome 15
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Unexposed Practice Group- Aim 1 | On-field Activity Group - Aim 3
Number analyzed (Participants) | 35 | 29
score on a scale | 0.37 (0.89) | 0.10 (0.39)

40. Secondary Outcome: Vestibular/Ocular Motor Screening (VOMS) - Vertical Saccades
Description: The participant will be asked to focus on two small targets that are vertically aligned, moving their eyes quickly from one target to the other. The participant will report any symptoms (i.e., headache, dizziness, nausea, fogginess) after the task is complete. Symptoms reported range on a scale from 0-10; lower scores are better.
Time Frame: Baseline
Population: as for outcome 15
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Unexposed Practice Group- Aim 1 | On-field Activity Group - Aim 3
Number analyzed (Participants) | 35 | 29
score on a scale | 0.34 (0.84) | 0.12 (0.36)

41. Secondary Outcome: Vestibular/Ocular Motor Screening (VOMS) - Vertical Saccades
Description: as for outcome 40
Time Frame: Month 3
Population: as for outcome 21
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Unexposed Practice Group- Aim 1 | On-field Activity Group - Aim 3
Number analyzed (Participants) | 25 | 21
score on a scale | 0.15 (0.49) | 0.10 (0.31)

42. Secondary Outcome: Vestibular/Ocular Motor Screening (VOMS) - Horizontal Vestibular Ocular Reflex
Description: The participant will be asked to focus on one small target while rotating their head from side to side. The participant will report any symptoms (i.e., headache, dizziness, nausea, fogginess) after the task is complete. Symptoms reported range on a scale from 0-10; lower scores are better.
Time Frame: Baseline
Population: as for outcome 15
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Unexposed Practice Group- Aim 1 | On-field Activity Group - Aim 3
Number analyzed (Participants) | 35 | 29
score on a scale | 0.29 (0.80) | 0.13 (0.36)

43. Secondary Outcome: Vestibular/Ocular Motor Screening (VOMS) - Visual Motion Sensitivity
Description: as for outcome 39
Time Frame: Month 3
Population: as for outcome 21
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Unexposed Practice Group- Aim 1 | On-field Activity Group - Aim 3
Number analyzed (Participants) | 25 | 21
score on a scale | 0.17 (0.52) | 0.10 (0.33)

44. Secondary Outcome: Vestibular/Ocular Motor Screening (VOMS) - Near Point Convergence
Description: The participant will be asked to focus on a small target and slowly bring it to the tip of their nose until two distinct images of the target are seen. The participant will complete this three times and scores will be averaged over three trials - Participants will complete a preseason baseline assessment which will be compared to post-season assessment scores - Rates changes in symptoms on 0 - 15; lower scores are better
Time Frame: Baseline
Population: as for outcome 15
Measure: Mean (Standard Deviation); unit: centimeters
Arm/Group | Unexposed Practice Group- Aim 1 | On-field Activity Group - Aim 3
Number analyzed (Participants) | 35 | 29
centimeters | 6.48 (5.71) | 2.97 (2.93)

45. Secondary Outcome: Vestibular/Ocular Motor Screening (VOMS) - Near Point Convergence
Description: as for outcome 44
Time Frame: Month 3
Population: as for outcome 21
Measure: Mean (Standard Deviation); unit: centimeters
Arm/Group | Unexposed Practice Group- Aim 1 | On-field Activity Group - Aim 3
Number analyzed (Participants) | 25 | 21
centimeters | 6.00 (4.92) | 3.38 (4.96)

46. Secondary Outcome: Conners' Continuous Performance Test (CPT) - Reaction Speed
Description: Participants will complete a 14-minute computer-based assessment that evaluates selective, sustained and divided attention, as well as impulsivity and vigilance - Participants will complete a preseason baseline assessment which will be compared to post-season assessment scores - CPT Reaction Speed; Raw reaction speed is the mean response speed for all non-perseverative responses made during the entire Test. Raw reaction speed is converted to standardized T-scores 0-90; 50 indicates the population mean with a standard deviation of 10. 70+ is atypically slow and <40 is atypically fast. Reaction speed is bi-directional with higher scores indicating slower reaction times (i.e., inattentiveness), and lower scores indicating faster reaction times (i.e., impulsivity)
Time Frame: Baseline
Population: Missing from each group-- Unexposed practice group: 1 incompatible with mouthpiece
  On-field activity group: 1 incompatible with mouthpiece, 1 received invalid CPT results, 1 didn't attend baseline testing, and 3 joined the study after the start of contact
Measure: Mean (Standard Deviation); unit: T-score
Arm/Group | Unexposed Practice Group- Aim 1 | On-field Activity Group - Aim 3
Number analyzed (Participants) | 35 | 28
T-score | 55.34 (11.77) | 47.00 (9.50)

47. Secondary Outcome: Conners' Continuous Performance Test (CPT)) - Omissions
Description: Participants will complete a 14-minute computer-based assessment that evaluates selective, sustained and divided attention, as well as impulsivity and vigilance - Participants will complete a preseason baseline assessment which will be compared to post-season assessment scores - CPT Omissions; Raw omissions scores are based on the number of missed targets during the test. Raw omissions scores are converted to standardized T-scores 0-90; 50 indicates the population mean with a standard deviation of 10. 70+ is very elevated and indicates poor performance. Higher scores indicate poorer performance
Time Frame: Baseline
Population: as for outcome 46
Measure: Mean (Standard Deviation); unit: T score
Arm/Group | Unexposed Practice Group- Aim 1 | On-field Activity Group - Aim 3
Number analyzed (Participants) | 35 | 28
T score | 64.46 (16.7) | 55.07 (14.99)

48. Secondary Outcome: Conners' Continuous Performance Test (CPT) - Omissions
Description: as for outcome 47
Time Frame: Month 3
Population: Missing participants--Unexposed group: 1 incompatible with mouthpiece, 1 had injury, 3 quit team, 1 did not like mouthpiece, 5 didn't return for post-season neurocognitive testing. On-field activity group: 1 incompatible with mouthpiece,1 athlete's parent withdrew consent, 4 quit the team, 2 didn't like mouthpiece, 1 received invalid CPT results, 1 did not attend baseline neurocognitive testing, 3 joined study after start of contact in season,1 athlete didn't return for post-season testing.
Measure: Mean (Standard Deviation); unit: T-score
Arm/Group | Unexposed Practice Group- Aim 1 | On-field Activity Group - Aim 3
Number analyzed (Participants) | 25 | 20
T-score | 61.68 (16.23) | 52.30 (12.04)

49. Secondary Outcome: Conners' Continuous Performance Test (CPT) - Commissions
Description: Participants will complete a 14-minute computerbased assessment that evaluates selective, sustained and divided attention, as well as impulsivity and vigilance - Participants will complete a preseason baseline assessment which will be compared to post-season assessment scores - CPT Commission; Raw commissions are incorrect responses to non-targets. Raw commissions scores are converted to standardized T-scores 0-90; 50 indicates the population mean with a standard deviation of 10. 70+ is very conservative and indicates much emphasis on accuracy over speed and ≤30 is very liberal and indicates much emphasis on speed over accuracy. Scores indicate the nature of participants' response style rather than performance
Time Frame: Baseline
Population: as for outcome 46
Measure: Mean (Standard Deviation); unit: T score
Arm/Group | Unexposed Practice Group- Aim 1 | On-field Activity Group - Aim 3
Number analyzed (Participants) | 35 | 28
T score | 52.57 (7.93) | 50.14 (8.15)

50. Secondary Outcome: Conners' Continuous Performance Test (CPT) - Commissions
Description: as for outcome 49
Time Frame: Month 3
Population: as for outcome 48
Measure: Mean (Standard Deviation); unit: T score
Arm/Group | Unexposed Practice Group- Aim 1 | On-field Activity Group - Aim 3
Number analyzed (Participants) | 25 | 20
T score | 50.56 (8.69) | 47.20 (8.82)

51. Secondary Outcome: Conners' Continuous Performance Test (CPT) - Perseverations
Description: Participants will complete a 14-minute computer-based assessment that evaluates selective, sustained and divided attention, as well as impulsivity and vigilance - Participants will complete a preseason baseline assessment which will be compared to post-season assessment scores - CPT Perseverations; Raw perseverations are responses that are made in less than 100 milliseconds following a stimulus. Raw perseverations scores are converted to standardized T-scores 0-90; 50 indicates the population mean with a standard deviation of 10. 70+ is very elevated and indicates poor performance. Higher scores indicate poorer performance
Time Frame: Baseline
Population: Missing participants-- Unexposed practice group: 1 incompatible with mouthpiece
  On-field activity group: 1 incompatible with mouthpiece, 1 received invalid CPT results, 1 didn't attend baseline testing, and 3 joined the study after the start of contact
Measure: Mean (Standard Deviation); unit: T score
Arm/Group | Unexposed Practice Group- Aim 1 | On-field Activity Group - Aim 3
Number analyzed (Participants) | 35 | 28
T score | 67.74 (18.71) | 58.00 (14.82)

52. Secondary Outcome: Conners' Continuous Performance Test (CPT) - Perseverations
Description: as for outcome 51
Time Frame: Month 3
Population: as for outcome 48
Measure: Mean (Standard Deviation); unit: T score
Arm/Group | Unexposed Practice Group- Aim 1 | On-field Activity Group - Aim 3
Number analyzed (Participants) | 25 | 20
T score | 68.48 (18.98) | 54.75 (16.46)

53. Secondary Outcome: Post Season (ImPACT) Immediate Post-Concussion Assessment and Cognitive Testing - Visual Motor Composite Score
Description: as for outcome 15
Time Frame: Month 3
Population: as for outcome 21
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Unexposed Practice Group- Aim 1 | On-field Activity Group - Aim 3
Number analyzed (Participants) | 25 | 21
score on a scale | 30.79 (7.48) | 30.30 (8.70)

54. Secondary Outcome: (ImPACT) Immediate Post-Concussion Assessment and Cognitive Testing - Reaction Time Composite Score
Description: as for outcome 18
Time Frame: Month 3
Population: as for outcome 21
Measure: Mean (Standard Deviation); unit: milliseconds
Arm/Group | Unexposed Practice Group- Aim 1 | On-field Activity Group - Aim 3
Number analyzed (Participants) | 25 | 21
milliseconds | 0.71 (0.12) | 0.70 (0.09)

55. Secondary Outcome: (ImPACT) Immediate Post-Concussion Assessment and Cognitive Testing - Impulse Control Composite Score
Description: as for outcome 19
Time Frame: Month 3
Population: as for outcome 21
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Unexposed Practice Group- Aim 1: Data from an unexposed sample (football players practicing as they would otherwise).
  These 11 athletes were excluded from month 3 neurocognitive data for the unexposed practice group
Arm/Group | Unexposed Practice Group- Aim 1 | On-field Activity Group - Aim 3
Number analyzed (Participants) | 25 | 21
score on a scale | 11.80 (9.65) | 12.1 (13.13)

56. Secondary Outcome: NIH Toolbox Pattern Comparison Test Score
Description: The Pattern Comparison Test is a measure of speed of processing, which typically improves steadily (time to complete task decreases) throughout childhood and adolescence, then begins to decline in adulthood, becoming much slower in older adults. As such, it is considered a "fluid ability" measure. Score range: 0-130
Time Frame: Baseline
Population: as for outcome 15
Measure: Mean (Standard Deviation); unit: number items correct
Arm/Group | Unexposed Practice Group- Aim 1 | On-field Activity Group - Aim 3
Number analyzed (Participants) | 35 | 29
number items correct | 91.03 (26.49) | 102.10 (26.3)

57. Secondary Outcome: NIH Toolbox Pattern Comparison Test Score
Description: as for outcome 56
Time Frame: Month 3
Population: as for outcome 21
Measure: Mean (Standard Deviation); unit: number items correct
Arm/Group | Unexposed Practice Group- Aim 1 | On-field Activity Group - Aim 3
Number analyzed (Participants) | 25 | 21
number items correct | 106.12 (19.78) | 113.86 (27.89)

58. Secondary Outcome: (ImPACT) Immediate Post-Concussion Assessment and Cognitive Testing - Verbal Memory Composite Score
Description: as for outcome 15
Time Frame: Month 3
Population: as for outcome 21
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Unexposed Practice Group- Aim 1 | On-field Activity Group - Aim 3
Number analyzed (Participants) | 25 | 21
score on a scale | 84.96 (10.98) | 81.62 (15.04)

59. Secondary Outcome: (ImPACT) Immediate Post-Concussion Assessment and Cognitive Testing - Visual Memory Composite Score
Description: as for outcome 15
Time Frame: Month 3
Population: as for outcome 21
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Unexposed Practice Group- Aim 1 | On-field Activity Group - Aim 3
Number analyzed (Participants) | 25 | 21
score on a scale | 73.76 (10.28) | 68.29 (16.35)

60. Secondary Outcome: Vestibular/Ocular Motor Screening (VOMS) - Horizontal Vestibular Ocular Reflex
Description: as for outcome 42
Time Frame: Month 3
Population: as for outcome 21
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Unexposed Practice Group- Aim 1 | On-field Activity Group - Aim 3
Number analyzed (Participants) | 25 | 21
score on a scale | 0.15 (0.46) | 0.10 (0.31)

61. Secondary Outcome: Conners' Continuous Performance Test (CPT) - Reaction Speed
Description: as for outcome 46
Time Frame: Month 3
Population: as for outcome 48
Measure: Mean (Standard Deviation); unit: T score
Arm/Group | Unexposed Practice Group- Aim 1 | On-field Activity Group - Aim 3
Number analyzed (Participants) | 25 | 20
T score | 51.48 (11.33) | 45.60 (4.42)

ADVERSE EVENTS:
Time Frame: 13 weeks
Description: Study team depended on Parents and Coaches to report AEs
Groups:
- Unexposed Practice Group- Aim 1 Stakeholders: Data from an unexposed sample
- On-field Activity Group - Aim 3 Stakeholders: participation in this research will involve 4 to 12 visits and last about 1 hour per meeting over 4 to12 months - Participation in this study will involve discussion of biomechanical and video data with other stakeholders via semi-structured focus groups (coaches and parents) or individual interviews with league officials surrounding awareness and receptivity to creating a safer practice structure
- Unexposed Practice Group - Other Stakeholders: : Parent and organizational leader stakeholders (unexposed to intervention) participated in guided discussions about safety and biomechanics in youth football
Arm/Group | Unexposed Practice Group- Aim 1 | On-field Activity Group - Aim 3 | Unexposed Practice Group- Aim 1 Stakeholders | On-field Activity Group - Aim 3 Stakeholders | Unexposed Practice Group - Other Stakeholders
All-Cause Mortality (participants affected / at risk) | 0/36 | 0/34 | 0/6 | 0/12 | 0/18
Serious Adverse Events (participants affected / at risk) | 0/36 | 0/34 | 0/6 | 0/12 | 0/18
Other Adverse Events (participants affected / at risk) | 0/36 | 0/34 | 0/6 | 0/12 | 0/18

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2024-08-21): https://cdn.clinicaltrials.gov/large-docs/30/NCT04908930/Prot_SAP_001.pdf
  • Informed Consent Form (2023-08-21): https://cdn.clinicaltrials.gov/large-docs/30/NCT04908930/ICF_000.pdf